CLINICAL TRIAL: NCT07091123
Title: Patient Preference and Long-term Outcomes in Persistent Spinal Pain Syndrome: A Prospective Study Comparing Spinal Cord Stimulation to Intrathecal Drug Delivery.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Salim M Hayek, Chief of the Division of Pain Medicine at University Hospitals, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY20241226
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Persistent Spinal Pain Syndrome
Keywords: Pain pump; neuromodulation prognostic tests
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group A (Active Comparator): SCS prognostic test performed first followed about 2-4 weeks later with continuous IDD test with bupivacaine 0.625 mg/ml and fentanyl 2 mcg/ml for 8-23 hours.
  Interventions: Device: Pain pump; Drug: Bupivacain 0.625%/Fentanyl 2mcg/ml; Device: Spinal Cord Stimulator (SCS)
- Group B (Active Comparator): IDD prognostic test for 8-23 hours followed 2-4 weeks later by SCS prognostic test.
  Interventions: Device: Pain pump; Drug: Bupivacain 0.625%/Fentanyl 2mcg/ml; Device: Spinal Cord Stimulator (SCS)

INTERVENTIONS:
Device: Pain pump — Spinal catheter place under local anesthesia.
Drug: Bupivacain 0.625%/Fentanyl 2mcg/ml — A solution containing fentanyl 2 mcg/mL and bupivacaine 0.625 mg/mL at an infusion rate of 0.5 ml/hr.
Device: Spinal Cord Stimulator (SCS) — Two spinal cord stimulation leads will then be advanced under fluoroscopy to the target area, typically around T7-T9 in the posterior epidural space.
  Currently, there are six manufacturers of spinal cord stimulation devices with implanted programmable generators or receivers.

SUMMARY:
Spinal cord stimulation (SCS) or intrathecal drug delivery (pain pump) can be effective in providing pain relief for patients with low back pain who have not responded to other treatments. While both treatments, SCS and pain pump, may help with low back pain relief, it is not known which treatment may work better for patients. SCS and pain pumps involve an implanted device in the body.

In this study, we are asking patients to undergo a trial of both treatment modalities, SCS and pain pump, as screening tests prior to considering an implant. A total of 36 patients will be enrolled in this study. After both trials are completed, participants will be seen in the office and asked which treatment modality they believe has been more effective for relieving pain during the trial periods by completing questionnaires. If neither treatment was effective in improving baseline pain by at least 50%, participants would not qualify for either implant whether or not they are part of this study. Direct study participation would end here. If either or both treatment modalities improved baseline pain by at least 50%, participants will be asked to choose the treatment that worked better: SCS or pain pump. Participants will then have the option to proceed to the permanent implant of choice: SCS or pain pump. Direct study participation would end here but participants will then be followed in the doctor's office after implant as is customary for usual clinical care. The study data collection will conclude when the screening tests are completed.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 years or greater
* Previous lumbar or thoracic spine surgery
* Intractable pain of trunk (more than limbs; ≥ 75%/25% ratio back/leg pain)
* Patient who passed psychological evaluations as part of the usual clinical care prior to consideration of IDDS and are stable with current pain condition and medications
* Failed more conservative management, including physical therapy, medications and injections.

Exclusion Criteria:

* Untreated infection or coagulopathy/patient unable to stop anticoagulants
* Immune compromised state precluding having an implant
* Allergic reactions to bupivacaine or fentanyl
* Pregnancy.
* Patients using > 15 mg oral equivalents of morphine daily or who are unable to wean down below that dosage for 4 weeks or more before the prognostic test date
* Neurological deficits characterized as weakness in lower extremities with evidence of nerve damage resulting in difficulty ambulating
* Patients deemed by Spine Surgery to be candidates for revision lumbar spine surgery

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2027-08-11 (Estimated); Study Completion 2027-08-11 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity as measured by Numerical Rating Scale [NRS] | Baseline, up to 23 hours after catheter placement (for IDD group) Baseline, one week after lead placement (for SCS group) 3, 6, 12 months for implanted patients
  Numerical Rating Scale [NRS] is a numbered scale, from 0 to 10, where 0 represents no pain and 10 represents the worst pain imaginable
Change in pain intensity as measured by Oswestry disability index [ODI] | Baseline, up to 23 hours after catheter placement (for IDD group) Baseline, one week after lead placement (for SCS group), 3, 6, 12 months for implanted patients
  Oswestry disability index [ODI] is a questionnaire used to assess the impact of low back pain on a person's daily life. The ODI score ranges from 0 to 100, with lower scores indicating less disability.
Change in pain intensity as measured by painDETECT | Baseline, up to 23 hours after catheter placement (for IDD group) Baseline, one week after lead placement (for SCS group), 3, 6, 12 months for implanted patients
  painDETECT is a nine-item questionnaire. A total score of 19 or more is indicative of likely neuropathic pain.

SECONDARY OUTCOMES:
Change in quality of life as measured by the PROMIS-29. | Baseline, up to 23 hours after catheter placement (for IDD group) Baseline, one week after lead placement (for SCS group), 3, 6, 12 months for implanted patients
  PROMIS-29 is 29 item patient reported outcome tool measuring health-related quality of life. With higher scores indicating higher quality of life.
Number of adverse events as measured by patient report, | Up to 12 months
Change in daily opioid consumption as measured by Rx report | 3, 6, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Salim Hayek, MD, Principal Investigator — University Hospitals
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No